CLINICAL TRIAL: NCT05538884
Title: A Novel Intertransverse Plane Block: A Magnetic Resonance Imaging and Volunteer Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Si 267/2022
Record Dates: First submitted 2022-09-11; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Intertransverse Process Block; Thoracic Nerve Block; Thoracic Paravertebral Block
Keywords: MRI study; Volunteer study

STUDY DESIGN:
Intervention Model Description: The ITPB block at T5-6 level will be performed with a mixture of local anesthetic with MRI contrast 0.5% bupivacaine 10 ml and 0.5 ml contrast in concentration 3.09 mmol/l. Volunteers will be moved to MRI machine and imaged in a supine position for their whole thoracic spine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intertransverse process block (Experimental): Using a simple transverse ultrasound imaging technique to visualize the superior costotransverse ligament (SCTL) and the retro-SCTL space, we can perform a novel ITPB. Local anesthetic will be injected at the retro SCTL space.
  Interventions: Procedure: Intertransverse process block

INTERVENTIONS:
Procedure: Intertransverse process block — The ITPB block at T5-6 will be performed with a mixture of local anesthetic with MRI contrast 0.5% bupivacaine 10 ml and 0.5 ml contrast in concentration 3.09 mmol/l. Volunteers will be moved to MRI machine and imaged in a supine position for their whole thoracic spine. This process will last about 45-60 minutes.

SUMMARY:
Intertransverse process block (ITPB) is a thoracic nerve block technique where the LA is injected into the thoracic "intertransverse tissue complex" posterior to the superior costotransverse ligament (SCTL). It may be an attractive alternative to a TPVB for unilateral surgery on the thorax, when considering the risk for pleural puncture, since it does not require direct needle access to the thoracic paravertebral space. However, although ITPB is ultrasound guided, the LA is frequently injected using surrogate bony landmarks in the sagittal sonogram, and in most cases without even identifying the SCTL.

DETAILED DESCRIPTION:
The knowledge regarding the spread of local anesthetic is a major prerequisite for a safe and effective use of all regional anesthetic methods in clinical practice. The primary outcome is the spread of injectate which will be evaluated on axial three-dimensional MRI with contrast medium. The secondary outcome is the sensory dermatomal blockade of this novel ITPB block.

ELIGIBILITY:
Inclusion Criteria:

* healthy Thai men with no diseases

Exclusion Criteria:

* inability to cooperate or communicate in Thai
* BMI ≥ 30 kg/m2 or body weight ≤ 45 kgs
* allergy to local anesthetics or contrast agents
* infection in the block area
* previous surgery or anatomical abnormalities of thoracic spines closed to block area
* coagulation disorder/thrombocytopenia/anticoagulation therapy
* contraindications to magnetic resonance imaging (MRI) (metal implants - pacemaker and others, claustrophobia)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Local anesthetic spreading from MRI image | 1 month
  Using local anesthetic mixed with contrast

CONTACTS AND LOCATIONS:
Overall Officials: Pawinee Pangthipampai, Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No